CLINICAL TRIAL: NCT00641420
Title: Safety and Efficacy of 1550nm Fractional Laser Treatment for Acne Scars in Fitzpatrick Type IV-VI Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David M. Ozog, Senior Staff, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HenryFord4447
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Acne Scarring
Keywords: Acne scarring; Post inflammatory hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fractional Laser 10mJ (Experimental): Patients receive fractional laser resurfacing to 17% of the face five times one month apart at 10mJ.
  Interventions: Procedure: Fractionated Laser Resurfacing
- Fractional Laser 40mJ (Experimental): Patients receive fractional laser resurfacing to 17% of the face five times one month apart at 40mJ.
  Interventions: Procedure: Fractionated Laser Resurfacing

INTERVENTIONS:
Procedure: Fractionated Laser Resurfacing
  Other Names: Fractionated Laser: FRAXEL

SUMMARY:
Fractionated laser resurfacing is commonly used as a treatment for acne scarring in fair skinned individuals. This study aims to test the efficacy and safety in darker skin types. Patients are randomized to either the 10mJ 40mJ dosages and receive a total of five treatments at 17% one month apart. Improvement is judged by a dermatologist as 0-25%, 25-50%, 50-75% or 75-100%. Side effects such as pigmentary abnormalities and pain are also evaluated.

DETAILED DESCRIPTION:
Background: Ablative resurfacing lasers are effective for treatment of acne scars, but they have a high risk of complications. Fractional lasers have less severe side effects but more moderate efficacy than ablative devices. Studies were performed in individuals with Fitzpatrick skin type I to VI.

Objective: To determine the efficacy and safety of an erbium 1,550-nm fractional laser in the treatment of facial acne scars in Fitzpatrick skin types IV to VI.

Methods: We conducted a prospective, single-blind, randomized trial in patients with acne scars (n=15), skin type IV to VI, with a 1,550-nm erbium fractionated laser. Patients were divided into two groups; one was treated with 10 mJ and the other with 40 mJ. Five monthly laser sessions were performed. A patient questionnaire was distributed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female voluntary patients between the ages of 18 and 59 with Fitzpatrick skin type IV-VI as verified by one of the investigators
* Patients with clinical diagnosis of ice pick, rolling, or boxcar type ane scarring
* Patients able to follow instructions
* If patient has a history of cold sores (herpes labialis) they must be willing to take prophylactic valtrex
* Written informed consent from the patients (Appendix II)

Exclusion Criteria:

* Children (less than 18 years old)
* Pregnant or lactating women
* Personal history of keloids or hypertrophic scarring
* Active acne requiring topical or oral therapy
* Accutane or other oral retinoid in past year
* Patients with a known allergy to lidocaine
* Allergy to valacyclovir in a patient that needs prophylaxis
* Patients with an unstable or non controlled underlying medical problem
* Patients who are not able to follow instructions
* Patients who have participated in a study within the 3 months prior to study entry
* Patients who refuse to give written informed consent
* Patients with a history of a pigmentary abnormality

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Improvement in acne scarring. | 6 months
  Blinded evaluators will score improvement of acne via photographs using a quartile grading scale (0 = no improvement, 1 = minor improvement [1-25%], 2 =moderate improvement [26-50%], 3 =marked improvement [51-75%], 4 = very significant improvement [76-100%]).

SECONDARY OUTCOMES:
Dyspigmentation | 6 months
  dyspigmentation will be assessed separately from acne scarring via photographs with blinded evaluators on a scale of 1- 3. 1 (minimal amount of hyperpigmentation), 2 (moderate hyperpigmentation) and 3 (severe amount of hyperpigmentation) depending on the degree of hyperpigmentation compared with their baseline photo.
Pain with treatment | 5 months
  subjects will report any pain with treatment on a 0-10 scale, with zero indicating no pain and 10 indicating the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: David M Ozog, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States